CLINICAL TRIAL: NCT04988113
Title: Presentation And Management Of Neglected Inhaled Foreign Body At Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Abdallah Mohamed Ahmed, resident, Sohag University
Other Study IDs: Soh-Med-21-07-14
Record Dates: First submitted 2021-07-13; First posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Foreign Body; Inhalation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Delayed presentation is not uncommon in children and may have been treated as asthma due to associated with low-grade cough and noisy breathing.

Late diagnoses of foreign body aspiration were defined as occurring beyond 3 days after the aspiration of the foreign body, or onset of symptoms.

Undiagnosed foreign body aspiration can cause mechanical effects, chemical reactions, and the most common complications were pneumonia, asthma, lung collapse, bronchiectasis, emphysema, mediastinal shift, atelectasis and lung abscess. Long-term presence of FBs in the bronchus may lead to bronchial stenosis

DETAILED DESCRIPTION:
A foreign body is an endogenous or exogenous substance, different from the anatomy of the site where it is found. Chevalier Jackson defined a foreign body as "an object or a substance that is foreign to its location".

Aspiration of a foreign body (FB) is a potentially life-threatening emergency and 75% of cases occur in children younger than 3 years of age, due to the absence of molar teeth, underdeveloped swallowing coordination and the tendency to talk and play while eating .

However, foreign body aspiration does happen in adults and elderly people as well.

Obtaining a good history plays a vital role in effectively diagnosing a foreign body aspiration. Three clinical phases of aspiration of foreign bodies are recognized: The first stage is the impaction of the foreign body and entitled "penetration syndrome," defined as a sudden onset of choking and intractable cough with or without vomiting.

In the second stage, these symptoms diminish as the foreign body settles into a stationary location and the tracheoesophageal reflexes tire out; this asymptomatic stage can last hours to weeks, which may delay diagnosis. In the third phase, Complications occur (also defined as Complications phase), when obstruction, erosion or infection cause pneumonia, atelectasis, abscess or fever. The first presentation of the condition may actually represent a complication of inhaled foreign body.

Delayed presentation is not uncommon in children and may have been treated as asthma due to associated with low-grade cough and noisy breathing.

Late diagnoses of foreign body aspiration were defined as occurring beyond 3 days after the aspiration of the foreign body, or onset of symptoms.

Undiagnosed foreign body aspiration can cause mechanical effects, chemical reactions, and the most common complications were pneumonia, asthma, lung collapse, bronchiectasis, emphysema, mediastinal shift, atelectasis and lung abscess. Long-term presence of FBs in the bronchus may lead to bronchial stenosis.

Neglected foreign bodies in the respiratory tract may occur due to misdiagnosis by the fellow professionals and pediatricians when FBs in the upper tracheal airway produce symptoms similar to those of viral subglottic croup or due to lack of typical symptoms and signs. The most common symptoms and signs of FBA, namely coughing, wheezing, and decreased air entry, can easily be overlooked by bronchial asthma or pneumonia. Parental negligence, not conclusive chest radiographs, and false negative bronchoscopic findings are other blamed factors

ELIGIBILITY:
Inclusion Criteria:

Patients who were diagnosed with neglected inhaled foreign body who underwent bronchoscopy in sohag university hospital, all ages, both Gender.

Exclusion Criteria:

Patients who were diagnosed with recent inhaled foreign body.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Patients who were diagnosed with neglected inhaled foreign body who underwent bronchoscopy in sohag university hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of different pictures of clinical presentations in neglected inhaled foreign body. | 3 months from August to December 2021
  This is a retrospective study that will be conducted in our tertiary center "Sohag University Hospital", will include cases of neglected inhaled foreign bodies in the period from June 2016 to June 2021, the medical records of patients who underwent bronchoscopy for suspected neglected foreign body aspiration will be reviewed. Assessment of different pictures of clinical presentations by reviewed symptoms and signs for the cases.
Determination of types of complications in neglected inhaled foreign body. | 3 months from August to December 2021
  This is a retrospective study that will be conducted in our tertiary center "Sohag University Hospital", will include cases of neglected inhaled foreign bodies in the period from June 2016 to June 2021, the medical records of patients who underwent bronchoscopy for suspected neglected foreign body aspiration will be reviewed. Determination of types of complications in neglected inhaled foreign body.
Determination of different types of management plans in neglected inhaled foreign body. | 3 months from August to December 2021
  This is a retrospective study that will be conducted in our tertiary center "Sohag University Hospital", will include cases of neglected inhaled foreign bodies in the period from June 2016 to June 2021, the medical records of patients who underwent bronchoscopy for suspected neglected foreign body aspiration will be reviewed. Determination of different types of management plans by rigid or flexible bronchoscopic findings, including the type and the location of the foreign body

CONTACTS AND LOCATIONS:
Overall Officials: Abdel-Mateen M Abd ElLateef, professor, Study Chair — Sohag University
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adjeso T, Damah MC, Murphy JP, Anyomih TTK. Foreign Body Aspiration in Northern Ghana: A Review of Pediatric Patients. Int J Otolaryngol. 2017;2017:1478795. doi: 10.1155/2017/1478795. Epub 2017 Oct 1. PMID 29098005
- [Background] Lin L, Lv L, Wang Y, Zha X, Tang F, Liu X. The clinical features of foreign body aspiration into the lower airway in geriatric patients. Clin Interv Aging. 2014 Sep 24;9:1613-8. doi: 10.2147/CIA.S70924. eCollection 2014. PMID 25284994
- [Background] Salih AM, Alfaki M, Alam-Elhuda DM. Airway foreign bodies: A critical review for a common pediatric emergency. World J Emerg Med. 2016;7(1):5-12. doi: 10.5847/wjem.j.1920-8642.2016.01.001. PMID 27006731